CLINICAL TRIAL: NCT01577498
Title: Age Estimation of Adolescents for Legal Purposes: Determining the Medical Response
Brief Title: Age Estimation of Adolescents for Legal Purposes
Acronym: AGE-ADO
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: AOR 11118
Record Dates: First submitted 2012-03-30; First posted 2012-04-13 (Estimated); Last update posted 2016-06-10 (Estimated); Status verified 2016-05

CONDITIONS: Adolescence; Bone Maturation
Keywords: Skeletal age; Chronological age; Adolescent

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Economic globalisation has been associated with a rise of cross-border migration in Europe. In France, courts commonly demand appropriate medical tests aimed at age estimations of supposed minors without documentation. Determining the age of foreign adolescents may be important in order to define the rights and protection afforded them by law depending on this status, and the conditions in which they may be detained or held in police custody if they are under suspicion. Age estimation is considered to be ideally based on the combination of clinical, skeletal, and dental examinations. A number of forensic physicians do not integrate published recommendations or the results of published studies into their daily practice. Previous studies have shown that medical practice is heterogeneous in this area. Factors determining this heterogeneity are unknown.

We hypothesize that the personal and professional development of the physician, as well as the characteristics and the circumstances of medical examination can affect medical response on age determination, beyond clinical and radiological data. The purpose of this study is to identify factors determining medical response to courts.

DETAILED DESCRIPTION:
Economic globalisation has been associated with a rise of cross-border migration in Europe. Courts commonly demand appropriate medical tests aimed at age estimations of supposed minors without documentation. Determining the age of foreign adolescents may be important in order to define the rights and protection afforded them by law depending on this status, and the conditions in which they may be detained or held in police custody if they are under suspicion.

Guidelines for age estimation in living individuals have been proposed and are based on the combination of general clinical, skeletal, and dental examinations. However, guidelines for paediatricians in the UK and a national consensus conference in France on doctors' attendance on detainees in police custody have stated that the currently available methods generally do not enable a doctor to state with confidence if a detainee is a minor or not. The validity of currently used methods has also been questioned by the French National Consultative Ethics Committee on Health and Life Sciences.

As any middle school teacher can testify, anthropometric measures such as height and weight, and visible signs of sexual maturity vary widely from one adolescent to another, so that general clinical examination has limited value for age estimation. The skeletal examination is considered more reliable. In the reference radiological method, X-ray examination of the left hand and wrist is compared with standard images from an atlas published by Greulich and Pyle, who collected standards obtained in the 1930's and 1940's from an American white middle-class population. The main criteria applied for dental age determination are the eruption and development of the third molars, based on external and X-ray examination.

Age estimation is considered to be ideally based on the combination of clinical, skeletal, and dental examinations. However, it is not easy to determine from available published series if the estimated age of a given individual is a precise age or a spectrum of possible ages, and in this case how broad is the proposed spectrum. Indeed, the information in the radiological atlas by Greulich and Pyle is statistical, not individual. The use of such data for forensic purposes has never been intended by the authors, nor validated. Moreover, the ethnic and socioeconomic characteristics of the adolescents examined today in Western Europe may differ largely from those presented in the atlas, as previously suggested. The role of ethnic factors in skeletal maturation has been repeatedly studied and gave conflicting results. In most series evaluating skeletal age in different populations, hand and wrist X-rays were obtained from healthy subjects or patients received for evaluation of trauma. The conclusions of these studies may not be validated, or at least should be considered cautiously, when extrapolating results to adolescents without documents involved in judicial procedures, who have heterogeneous and largely unevaluated psychological and socioeconomic characteristics. A number of forensic physicians do not integrate published recommendations or the results of published studies into their daily practice. Previous studies have shown that medical practice is heterogeneous in this area. Factors determining this heterogeneity are unknown.

We hypothesize that the personal and professional development of the physician, as well as the characteristics and the circumstances of medical examination can affect medical response on age determination, beyond clinical and radiological data. The main objective of this study is to identify factors determining medical response to courts. A secondary objective is to evaluate how evidence-based data obtained from medical journals are taken into account in medical decision making by forensic physicians.

The main evaluated criterium is the medical response transmitted to courts regarding age determination.

Methods Prospective observational study of 500 age determinations requested by courts in migrant adolescents without documentation, in 18 departments of forensic medicine in France. Non-inclusion criterium is the refusal of the adolescent to undergo a medical examination.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent or young adult referred by judicial authorities for age determination

Exclusion Criteria:

* Refusal to undergo a medical examination

Ages: 10 Years to 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Adolescents or young adult addressed by the judicial police officer,for age determination in one of the participating centers
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2012-05; Primary Completion 2013-04 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Medical response transmitted to courts regarding age determination, at the end of medical examination | One hour

SECONDARY OUTCOMES:
Age evaluation based on published evidence on age determination, as evaluated by independent experts at 12 months | 12 months
  In each case, compatibility of (1) age (or age interval) transmitted to courts and (2) age evaluation based on published evidence on age determination, as evaluated by independent experts.

CONTACTS AND LOCATIONS:
Overall Officials: PATRICK CHARIOT, MD, Principal Investigator — AP-HP Hospital Jean Verdier
Locations (1):
- : Jean Verdier hospital, Department of forensic medicine, Bondy, France

REFERENCES:
- [Background] Pruvost MO, Boraud C, Chariot P. Skeletal age determination in adolescents involved in judicial procedures: from evidence-based principles to medical practice. J Med Ethics. 2010 Feb;36(2):71-4. doi: 10.1136/jme.2009.031948. PMID 20133398
- [Background] Buken B, Safak AA, Yazici B, Buken E, Mayda AS. Is the assessment of bone age by the Greulich-Pyle method reliable at forensic age estimation for Turkish children? Forensic Sci Int. 2007 Dec 20;173(2-3):146-53. doi: 10.1016/j.forsciint.2007.02.023. Epub 2007 Mar 27. PMID 17391883
- [Background] Schmeling A, Olze A, Reisinger W, Geserick G. Age estimation of living people undergoing criminal proceedings. Lancet. 2001 Jul 14;358(9276):89-90. doi: 10.1016/S0140-6736(01)05379-X. No abstract available. PMID 11463408
- [Background] Garamendi PM, Landa MI, Ballesteros J, Solano MA. Reliability of the methods applied to assess age minority in living subjects around 18 years old. A survey on a Moroccan origin population. Forensic Sci Int. 2005 Nov 10;154(1):3-12. doi: 10.1016/j.forsciint.2004.08.018. Epub 2004 Nov 10. PMID 16182943
- [Background] Hassanali J. The third permanent molar eruption in Kenyan Africans and Asians. Ann Hum Biol. 1985 Nov-Dec;12(6):517-23. doi: 10.1080/03014468500008091. PMID 4091506